CLINICAL TRIAL: NCT06587360
Title: Protocol for a Realist Evaluation and Feasibility RCT: Understanding and Developing a SPIKES-based eLearning Training Course Called fertiShare to Support Sharing Bad News Encounters Between Fertility Healthcare Professionals (FHPs) and Patients
Brief Title: fertiShare Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Wales Fertility Institute, Swansea Bay University Healthboard, Wales, UK (Unknown); Dept of Health Sciences, Milan University, Milan, Italy (Unknown)
Responsible Party: Principal Investigator, Sofia Gameiro, Principal Investigator, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SPON1955-23
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-12

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: sharing bad news; healthcare communication; assisted reproduction; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fertility Healthcare Provides (FHPs) will be randomised on a 1:1 ratio via computer-generated randomisation to have access to the fertiShare eLearning or a control condition eLearning (basic communication training), via a URL. Only the creative company responsible for the technical development of fertiShare know which URL (URL a or b) provide access to fertiShare and the control eLearnings. No trial participant (FHPs, patients), clinic managers and/or gatekeepers will be informed of the randomisation result. The trial management team (SG, JB) will know if participants were allocated to URL a or b. The data analyst will not know any randomisation result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fertiShare intervention (Experimental): sharing bad news eLearning course
  Interventions: Other: fertiShare intervention - sharing bad news eLearning course
- fertiShare control (Active Comparator): basic communication training skills eLearning course
  Interventions: Other: fertiShare control - basic communication skills eLearning course

INTERVENTIONS:
Other: fertiShare intervention - sharing bad news eLearning course — two-hour self-led eLearning course to support fertility staff in sharing bad news (SBN) with their patients
  organised in three modules. Module 1 explores definitions of bad news, why it is challenging to FHPs and patients, and the benefits of training. Module 2 offers SPIKES-based step-by-step guidance to ease SBNs. Module 3 offers guidance to cope with common challenges FHPs face: sharing bad news remotely, managing anger and uncertainty, and using good news to lessen the impact of bad news.
  Each module offers video content-based lessons, case studies that illustrate guidance and brief quizzes for self-reflection and assessment. Case studies show learners optimal and suboptimal approaches to SBN.
  Arms: fertiShare intervention
Other: fertiShare control - basic communication skills eLearning course — self-led eLearning course branded as fertiShare but designed to emulate the basic communication training healthcare providers receive as they undergo their professional degrees.
  organised in three modules. Module 1 explores definitions of bad news, why it is challenging to FHPs and patients, and the benefits of training. Module 2 introduces the communication cycle and associated communication techniques. Module 3 offers guidance regarding other basic communication skills: empathic communication, non-verbal communication, active listening and remote consultations, and communicating the likelihood of positive or negative treatment outcomes.
  Each module offers video content-based lessons, case studies, and brief quizzes. All teaching elements remain at the basic level (remembering and understanding instead of analysing and applying).
  Arms: fertiShare control

SUMMARY:
Sharing bad news (SBN) is a daily challenge for fertility staff and patients. Bad news happens at all stages of fertility care and includes e.g., diagnosing infertility, reporting unexpected, repeated, or definitive treatment failure. Extensive evidence shows that SBN triggers stress in staff due to anticipation of negative emotions and evaluations or, in extreme cases, even complaints and lawsuits. Inability to manage bad news can increase negative emotions in patients and fuel distrust, potentially leading to treatment discontinuation. Efficient SBN training exists but does not address challenges of SBN in fertility care, does not meet fertility staff training and patient care preferences, and its impact on patients is unclear.

fertiShare is a brief, evidence-based, e-Learning SBN course bespoke for fertility care. The aim of the study is to evaluate the feasibility of implementing fertiShare at fertility clinics and of implementing an online multi-centre RCT to determine fertiShare's efficacy. This will allow to conclude if fertiShare should proceed to efficacy evaluation.

An international interdisciplinary stakeholder group (patients, consultants, embryologists, nurses, psychologists, digital educators) will inform all aspects of the proposed project.

DETAILED DESCRIPTION:
The aim of the feasibility study is to make a fully informed decision about whether fertiShare should proceed to efficacy evaluation. This aim will be achieved by resolving uncertainties about implementing fertiShare at fertility clinics and about running an online multi-centre efficacy RCT for fertiShare.

Design: Pre-registered, online, multi-centre, two-arm, triple-blinded (staff, patients, data analysts), feasibility RCT with 1:1 computer-generated randomized allocation to the intervention (fertiShare) or minimal SBN information control (20 mins SBN lecture emulating what most staff would receive as part of general training) groups.

The trial will include a process evaluation and adopt a pragmatic attitude to maximise the applicability of findings to fertility care practice (beyond the immediate trial setting). Examples of design choices that translate this pragmatic attitude are our choice of the control condition (emulating general SBN training that most staff will have), the inclusion of multiple staff and patient secondary trial outcomes (informed by stakeholders) and low standardisation of intervention delivery (staff will apply fertiShare as they think best). Criteria for progression to efficacy evaluation will be specified prior to implementation using a traffic-light system.

Setting: Six UK-based private and public fertility clinics.

Participants: Staff working at clinics whose role involves 10% of week time SBN. Exclusion criteria are being unable to undergo training.

Patient inclusion criteria are having received bad news from participating staff within last month. No exclusion criteria are applied.

Bad news is defined as any news meaning that patients' first or second complete (fresh and frozen embryo transfers) initiated In Vitro Fertilization cycle did not result in a clinical pregnancy, as this is the most common challenging bad news shared by staff, and to ensure that patient outcome data (specifically continuation data) are comparable.

Guidance for feasibility studies to estimate participation rates, based on review of evidence from RCTs conducted within SBN training and fertility care, indicates 75% of staff will be eligible and participate, but a conservative estimate of 50% will be considered to decrease unknown risk. Recruiting 60 staff (10 per clinic) will allow to calculate a 50% participation rate to 95%CI of ±11%. 52% of patients will be eligible and participate. Recruiting 180 patients per cohort (30 per clinic) will allow to calculate a 60% participation rate to 95%CI of ±6%.

ELIGIBILITY:
Fertility Healthcare Professionals' inclusion criteria are:

* working at participating clinics; and
* whose role involves a minimum of 10% of week time (half a day) SBN or being a non-clinical decision-maker (e.g., clinic/line managers).

Patients' inclusion criteria are

• adult individuals or couples attending participating clinics to discuss or undergo (in)fertility diagnosis or treatment with participating FHPs.

Exclusion criteria are:

* not being able to read, speak or understand English;
* not being able to provide consent.
* for FHPs only, being unable to undergo the fertiShare training (e.g., visual impairments).

We will not be targeting groups or individuals deemed vulnerable. Potential participants are explicitly informed in the information sheet that, if they are worried about their mental health or psychological wellbeing they may chose not to participate at all. They are also advised to inform their fertility team and contact their GP in the usual way or the NHS Mental Health support service, www.nhs.yj/mental-health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Limited Efficacy Testing: changes from baseline in patients perceived FHPs' sharing bad news performance (primary outcome) | Within one week of enrolment in the study
  Modified intention-to-treat (mITT, all FHPs randomized) and per protocol (PP, only FHPs who completed a sufficient dose) analyses of mean differences in patient reported FHPs' sharing bad news performance (primary outcome) between patients in the baseline (pre FHPs training) and follow-up (post FHPs training) cohort. Patient reported FHPs' sharing bad news performance will be assessed with an adapted version of the Sharing Bad News Behavioural Assessment Scale. The scale is composed of 23 items that list evidence-based best practice behaviours on how to share bad news (e.g., warn you they would be sharing bad news). Patients are asked to rate the degree to which the FHP did each behaviour on a Likert scale from 1- not at all to 5 - completely (or 6 - does not apply). A global average score is calculated that ranges from 1 to 5, with higher values indicating better sharing bad news performance.

SECONDARY OUTCOMES:
Limited Efficacy Testing: changes from baseline in staff confidence in sharing bad news (secondary outcome) | From two weeks after enrolment to two weeks after training (fertiShare, control), which happens 5 months from enrolment
  Modified intention-to-treat (mITT, all FHPs randomized) and per protocol (PP, only FHPs who completed a sufficient dose) analyses of changes in confidence in SBN (secondary outcome) from pre to post training with fertiShare or control eLearning. Confidence in sharing bad news will be assessed with an adapted version of the Breaking Bad News Assessment Scale. The scale is composed of 23 items that list evidence-based best practice behaviours on how to share bad news (e.g., warn patients you will be sharing bad news). FHPs are asked to rate how confident they feel doing each behaviour listed on a Likert scale from 1- not at all to 5 - completely (or 6 - does not apply). A global average score is calculated that ranges from 1 to 5, with higher values indicating higher confidence in sharing bad news.
Limited Efficacy Testing: mean difference in patient trust in their Fertility Healthcare Professional (FHP) between the baseline and follow-up patient cohorts (secondary outcome) | Within one week of enrolment in the study
  Modified intention-to-treat (mITT, all FHPs randomized) and per protocol (PP, only FHPs who completed a sufficient dose) analyses of mean differences in patient trust in their FHP (secondary outcome) between patients in the baseline and follow-up cohort. Trust will be assessed with the Wake Forest Physician Trust Scale. The scale is composed of ten statements describing care provided (e.g., They will do whatever it takes to get you all the care you need.). Patients are asked to rate their level of agreement with each statement on a Likert scale from 1- strongly disagree to 5-strongly agree. Trust is measured by the sum of the 10 item scores (reverse-scored for negative items), ranging from 10 to 50, with a higher score indicating more trust.
Limited Efficacy Testing: mean difference in patients' satisfaction with care at the clinic (secondary outcome) between the baseline and follow-up patient cohorts | Within one week of enrolment in the study
  Modified intention-to-treat (mITT, all FHPs randomized) and per protocol (PP, only FHPs who completed a sufficient dose) analyses of mean differences in patient satisfaction with care at the clinic (secondary outcome) between patients in the baseline and follow-up cohort. Assessed with five questions used by the Human Fertility and Embryology Authority for patients to rate their satisfaction with care provided at UK based fertility clinics (e.g., To what extent did you feel you were treated with privacy and dignity?). Patients answer on a Likert scale from 1-never to 5-always (answer scale anchors vary with question), with higher values indicating higher satisfaction with care.
Limited Efficacy Testing: mean difference in patients' satisfaction with shared decision-making support regarding continuing or stopping fertility treatment (secondary outcome) between the baseline and follow-up patient cohorts (secondary outcome) | Within one week of enrolment in the study
  Modified intention-to-treat (mITT, all FHPs randomized) and per protocol (PP, only FHPs who completed a sufficient dose) analyses of mean differences in patient satisfaction with shared decision-making support about continuing fertility treatment (secondary outcome) between patients in the baseline and follow-up cohort. Assessed with the Decisional Conflict Scale. Patients are asked to select which treatment option they prefer (doing another treatment cycle at clinic, doing another treatment cycle at a different clinic, stopping fertility treatment, other) and to rate the degree to which they agree with a list of 16 statements related to their decision (e.g., I know which options are available to me) on a Likert scale from 0-strongly agree to 4-strongly disagree. Total decisional conflict and sub-dimension scores (uncertainty, informed, values clarity, support) are calculated and linearly transformed to range from 0 to 100, with higher scores indicating more of the construct.
Limited Efficacy Testing: mean difference in patients' uptake of and time to another stimulated In Vitro Fertilisation Cycle between the baseline and follow-up patients cohorts (secondary outcome) | 6 months and 2 weeks after enrolment
  Modified intention-to-treat (mITT, all staff randomized) and per protocol (PP, only staff who completed a sufficient dose) analysis of mean differences in patient uptake of (yes, no, not recommended) and time to another stimulated IVF cycle (in days, not applicable) between patients in the baseline and follow-up cohort: data obtained via patient record review.

OTHER OUTCOMES:
Demand of intervention: Fertility Healthcare Professionals demand for intervention | Within two weeks after exposure (fertiShare, control training), which happens 5 months from enrolment
  Number of Fertility Healthcare Professionals who registered with the eLearning and completed each lesson. module, and quiz
Demand for intervention: Profile of Fertility Healthcare Processionals who registered and completed the intervention | Within two weeks after exposure (fertiShare, control training), which happens 5 months from enrolment
  Demographic and professional profile of FHPs who registered and completed the intervention (fertiShare, control training)
Acceptability of intervention: Fertility Healthcare Professionals experience of doing intervention | Within two weeks after exposure (fertiShare, control training), which happens at 5 months from enrolment
  Quantitative ratings regarding 5 items describing the experience of doing the eLearning (e.g., I benefited, I learned). FHPs answer on a Likert-type scale ranging from 1 (not at all) to 5 (an extreme amount), presented in the eLearning evaluation form. Higher scores indicate higher acceptability of intervention.
Acceptability of intervention: Proportion of Fertility Healthcare Professionals recommending the intervention to colleagues | Within two weeks after exposure (fertiShare, control training), which happens at 5 months from enrolment
  Proportion of staff reporting they recommend fertiShare to other colleagues in their situation, fertiShare improved their preparation to have difficult conversations with their patients, and fertiShare reduced their anxiety when having difficult conversations with their patients: post-exposure (fertiShare, control training) staff assessment
Acceptability of intervention: patients' satisfaction with how their Fertility Healthcare Professional shared bad news with them | Within one week of enrolment in the study
  Patient self-reported satisfaction with how their FHP shared the bad news with them. Assessed with a single question "Overall, how satisfied are you with the way [name of participating staff member] shared or discussed with you the news that the IVF cycle was unsuccessful?", with a Likert-type response scale ranging from 1 (very dissatisfied) to 5 (very satisfied), presented in the patient pre- and post-cohorts' assessments
Acceptability of intervention: process evaluation interviews with Fertility Healthcare Professionals and patients | Within one to three months after exposure, which happens six to eight months after enrolment for FHPs and one month after for patients
  Open ended questions included in semi-structured process evaluation interviews with staff (e.g., Which aspects of FertiShare were particularly useful, if any?) and patients (e.g., What are your views about how staff shared with you the news that the IVF cycle was unsuccessful?)
Implementation of intervention: Number of Fertility Healthcare Professionals who completed all intervention (fertiShare, control training) Modules and completed Module 1 and 2 only during the 4-week training period | Within two weeks after exposure (fertiShare, control training), which happens at 5 months from enrolment
  Number of Fertility Healthcare Professionals who completed all intervention (fertiShare, control training) Modules (i.e., used intervention as intended) and completed Module 1 and 2 only (i.e., completed sufficient dose) during the 4-week training period: data stored by the eLearning
Implementation of intervention: process evaluation interviews with Fertility Healthcare Professionals and patients | Within one to three months after exposure, which happens six to eight months after enrolment for FHPs and one month after for patients
  Open ended questions included in semi-structured process evaluation interviews with FHPs (e.g., Can you describe any changes you made in the way you SBN with your patients (if any) because of doing the fertiShare eLearning and why?) and patients (e.g., Can you think of any factors that made it harder or easier for staff to share the news with you in a sensitive way?)
Practicality of intervention: Technical issues experienced by Fertility Healthcare Professionals | Within two weeks after exposure (fertiShare, control training), which happens at 5 months from enrolment
  Fertility Healthcare Professionals' answers to multiple choice question (yes, no) about experiencing technical issues during the intervention (fertiShare, control training), presented in the intervention Evaluation form
Practicality of intervention: process evaluation interviews with Fertility Healthcare Professionals and patients | Within one to three months after exposure, which happens six to eight months after enrolment for FHPs and one month after for patients
  Open ended questions included in semi-structured process evaluation interviews with FHPs (e.g., Where there any factors that made it easier or harder for you to do fertiShare?) and patients (e.g., Can you think of any factors that made it harder or easier for staff to share the news with you in a sensitive way?)
Demand of study protocol - Participation | Participation assessed at enrolment
  FHPs' and patients' participation (proportion of invited FHPs and patients who consent to participate) rates
Demand of study protocol - Retention | Retention assessment happens from 2 weeks to 5 months from enrolment for FHPs and within 2 weeks of enrolment for patients
  FHPs' and patients' retention rates (proportion of FHPs and patients who fill each assessment).
Acceptability of study protocol - Patients | Within two weeks of enrolment
  Proportion of patients in the pre- and post-training cohorts who complete their respective online assessments
Acceptability of study protocol - Fertility Healthcare Professionals | Within two weeks from enrolment and within two weeks after exposure, which happens 5 months from enrolment
  Proportion of FHPs who completed background and professional form, and pre- and post- exposure (fertiShare, control training) assessments
Implementation of study protocol | Fertility Healthcare Professionals: from enrolment until end of participation (seven months from enrolment). Patients: from enrolment until end of participation (within 2 weeks of enrolment).
  Issues reported by FHPs and patients to research team relating to study procedures or materials and reasons for non-participation/withdrawal from the study
Practicality of study protocol - Fertility Healthcare Professionals and Patients | Fertility Healthcare Professionals: At enrolment, within five, six and seven months of enrolment. Patients: At enrolment, within two weeks and two months of enrolment.
  Time taken by FHPs and patients to complete assessments and process evaluation interview
All dimensions - Process Evaluation Interviews | Fertility Healthcare Professionals: Withing 7 months of enrolment. Patients: within 2 months of enrolment.
  Open-ended questions included in semi-structured process evaluation interviews with FHPs and patients about the study methods (e.g., 'How demanding was participation in this study?' and, for staff only, 'How did you find the randomization process?')

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Gameiro, PhD, Principal Investigator — Cardiff University; Helen Falconer, Study Chair — Cardiff University
Locations (5):
- United Kingdom (5):
  - Aberdeen Fertility Centre, Aberdeen, Aberdeen
  - King's Fertility, London, London
  - Saint Mary's Hospital Manchester, Manchester University NHS Foundation Trust, Manchester, Manchester
  - The Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle, Newcastle upon Tyne
  - Wales Fertility Institute, Port Talbot, Port Talbot

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be submitted for publication. We will make the study data open on the Open Science Framework (with the participants' consent). This is an academic resource that makes data available for secondary analysis by other researchers and provides assurance of for science integrity and reproducibility.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start date: 01.01.2026, no end date.
URL: https://osf.io/9db52/

REFERENCES:
- [Background] Gameiro S, Adcock E, Graterol Munoz C, O'Hanrahan M, D'Angelo A, Boivin J. What is bad news in fertility care? A qualitative analysis of staff and patients' accounts of bad and challenging news in fertility care. Hum Reprod. 2024 Jan 5;39(1):139-146. doi: 10.1093/humrep/dead231. PMID 37968233
- [Background] Yilmaz Y, Sarikaya O, Senol Y, Baykan Z, Karaca O, Demiral Yilmaz N, Altintas L, Onan A, Sayek I. RE-AIMing COVID-19 online learning for medical students: a massive open online course evaluation. BMC Med Educ. 2021 May 27;21(1):303. doi: 10.1186/s12909-021-02751-3. PMID 34039344
- [Background] Miller SJ, Hope T, Talbot DC. The development of a structured rating schedule (the BAS) to assess skills in breaking bad news. Br J Cancer. 1999 May;80(5-6):792-800. doi: 10.1038/sj.bjc.6690423. PMID 10360657
- [Background] Hall MA, Zheng B, Dugan E, Camacho F, Kidd KE, Mishra A, Balkrishnan R. Measuring patients' trust in their primary care providers. Med Care Res Rev. 2002 Sep;59(3):293-318. doi: 10.1177/1077558702059003004. PMID 12205830
- [Background] Axboe MK, Christensen KS, Kofoed PE, Ammentorp J. Development and validation of a self-efficacy questionnaire (SE-12) measuring the clinical communication skills of health care professionals. BMC Med Educ. 2016 Oct 18;16(1):272. doi: 10.1186/s12909-016-0798-7. PMID 27756291
- [Derived] Gameiro S, Leone D, D'Angelo A, Veleva Z, Morey R, Boivin J. Multicentre pragmatic randomised controlled feasibility trial of fertiShare, a brief eLearning course to increase fertility staff performance when sharing bad news with their patients - a protocol. BMJ Open. 2025 Aug 25;15(8):e101269. doi: 10.1136/bmjopen-2025-101269. PMID 40854842